CLINICAL TRIAL: NCT05715281
Title: Rapid Analysis and Response Evaluation of Combination Anti-Neoplastic Agents in Rare Tumors (RARE CANCER) Trial: RARE 3 Tiragolumab + Atezolizumab
Brief Title: Testing the Combination of Anti-cancer Drugs Atezolizumab and Tiragolumab in People With Advanced Stage Rare Cancers, RARE3 Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-00705; NCI-2023-00705 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB001590; 10561 (Other: National Cancer Institute LAO); 10561 (Other: CTEP)
Record Dates: First submitted 2023-02-04; First posted 2023-02-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Rare Malignant Solid Neoplasm; Rare Malignant Solid Neoplasm; Refractory Rare Malignant Solid Neoplasm
MeSH Terms: interventions — atezolizumab; Biopsy; Specimen Handling; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (atezolizumab, tiragolumab) (Experimental): Patients receive atezolizumab IV over 60 minutes and tiragolumab IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO at baseline, undergo biopsy at baseline and on study, and undergo CT and collection of blood samples throughout the study.
  Interventions: Biological: Atezolizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Tiragolumab

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Tiragolumab — Given IV

SUMMARY:
This phase II trial tests how well atezolizumab works in combination with tiragolumab in treating patients with rare solid tumors that may have spread from where they first started to nearby tissue, lymph nodes, or distant parts of the body (advanced stage). Immunotherapy with monoclonal antibodies, such as atezolizumab and tiragolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The study biopsy takes small pieces of cancer tissue from a tumor. The purpose of these biopsies is to compare the body's immune response against the tumor before and after treatment with the study drugs. Blood samples will also be collected for the study. The researchers will use the samples to learn more about how atezolizumab and tiragolumab work and which patients in the future might be most likely to respond to atezolizumab and tiragolumab. Using atezolizumab in combination with tiragolumab may help to shrink tumors in patients diagnosed with advanced stage rare solid-tumor cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the proportion of activated CD8+ T cells at baseline and after treatment with atezolizumab and tiragolumab.

SECONDARY OBJECTIVES:

I. Determine the objective response rate (ORR) of patients with advanced rare cancers to the combination of atezolizumab and tiragolumab using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 and Immune-Modified (i)RECIST guidelines.

II. Measure progression-free survival (PFS) time (time frame: baseline until disease progression, death, loss to follow-up, initiation of another anti-cancer treatment, withdrawal of consent, or study termination).

III. Measure the proportion of patients with a clinically promising increase in CD8+ T cell infiltration following treatment with atezolizumab and tiragolumab.

EXPLORATORY OBJECTIVES:

I. Investigate immune activation markers and the immune composition (regulatory T [Treg], natural killer [NK], B-cells, macrophages, myeloid-derived suppressor cells [MDSC], tumor mutation burden [TMB], microsatellite instability [MSI]) in tumor microenvironment (TME) before and after study treatment.

II. Measure T cell receptor (TCR) signaling in tumor-infiltrating T cells in the TME as well as in circulating T cells in blood before and after study treatment using multiplex immunofluorescence assays (IFAs)-developed by the National Cancer Institute (NCI)-Frederick Pharmacodynamic Assay Development & Implementation Section (PADIS)-and use these measurements to evaluate the relationship between TCR signaling in circulating T cells and TME.

III. Evaluate potential associations between atezolizumab and tiragolumab activity and tumor genomic alterations, genomic expression, or TMB as determined from genomic analysis of biopsy samples.

IV. Evaluate genomic alterations in cell free deoxyribonucleic acid (DNA) (cfDNA) and their potential association with therapy response or resistance.

V. Evaluate the pharmacodynamic effects of the treatment on biomarkers of cell death and epithelial-to-mesenchymal transition (EMT) in tumor tissue and circulating tumor cells (CTCs).

VI. Evaluate markers of immune response and the presence of tertiary lymphoid structures (TLS) in TME at baseline and following atezolizumab plus tiragolumab therapy.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 60 minutes and tiragolumab IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) at baseline, undergo biopsy at baseline and on study, and undergo computed tomography (CT) and collection of blood samples throughout the study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed rare solid tumors that have progressed on standard therapy or for whom there is no standard of care therapy

  * Patients must not be eligible for a higher priority study that would be feasible for them to enroll in, such as a disease specific study of phase 2 or higher or a randomized study. Specifically, patients who are eligible for the PEP-CTN pediatric trial of atezolizumab and tiragolumab in children, adolescents, and young adults with SMARCB1- or SMARCA4-deficient tumors should be excluded
* Patients must have measurable disease as defined by RECIST v1.1, with at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam)
* Patients must have a tumor site amenable to biopsy
* Age >= 18 years. Because biopsies are mandatory on this trial, patients < 18 years of age are excluded
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* International normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 institutional upper limit of normal (ULN)

  * Patients who receive therapeutic anticoagulation therapy should be on a stable dose
* Total bilirubin =< 1.5 x institutional ULN (however, patients with known Gilbert disease who have serum bilirubin level of up to 3 mg/dl may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Creatinine =< 1.5 x institutional ULN OR creatinine clearance levels >= 30 mL/min/1.73 m^2 are permitted as the study agents are not secreted by the kidney
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for more than >= 1 month after treatment of the brain metastases
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Willingness to provide biopsy samples for research purposes
* Administration of atezolizumab and tiragolumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior monoclonal antibody therapy must have completed that therapy >= 5 weeks (or 3 half-lives of the antibody, whichever is shorter) prior to start of treatment (minimum of 1 week between prior therapy and study enrollment)
* Patients must have recovered from clinically-significant adverse events of their most recent cancer immunotherapy to grade 1 or less, (with the exception of alopecia and lymphopenia)
* Patients who are receiving any other investigational agents
* Prior anti-TIGIT therapy is not allowed. However, other prior immune checkpoint inhibitor therapy is permitted
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies (i.e., antibodies with generic names ending in "ximab" or "zumab", respectively) or fusion proteins, not resolved by pre-medication or steroids, leading to subsequent treatment cessation. Patients with a history of allergic reaction to chimeric or humanized antibodies for which symptoms never recurred after subsequent re-challenge may be considered after careful medical history review
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone [> 10 mg/day], cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and systemic mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients with uncontrolled intercurrent illness, that would limit compliance with study requirements
* Pregnant women are excluded from this study because atezolizumab and tiragolumab are investigational agents with unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, and because it is not known if tiragolumab can be excreted in human milk, breastfeeding should be discontinued if the mother is treated with atezolizumab
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with autoimmune hyperthyroid disease not requiring immunosuppressive treatment may be eligible
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Patients who have undergone major surgical procedures prior to Cycle 1, Day 1 who have not recovered to ECOG performance status =< 2 (Karnofsky >= 60%)
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to Cycle 1, Day 1 or at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of active CD8+ T cells infiltrating the tumor | At baseline and beginning of cycle 3
Pharmacodynamic (PD) response rate | At baseline, end of cycle 3, then every 2-4 cycles until disease progression
  The proportion of patients with a clinically promising increase in CD8+ T cell infiltration, defined as more than 1.5 standard deviations (SD) (as measured at baseline).
Incidence of adverse events | Cycle 1 day 1 to 30 days after last dose
  Reported using the common terminology criteria for adverse events version 5.0.

SECONDARY OUTCOMES:
Objective tumor response rate (ORR) | Up to 2 years
  Fifteen enrolled patients will yield 10 patients with evaluable paired biopsies with .95 probability, yielding 88% power, at the 1-sided .05 significance level, to detect an increase more than 1.25 SD (as measured at baseline), and to declare the combination promising with respect to the primary PD endpoint. This number will also be sufficient for assessment of the secondary endpoint of ORR; there will be 96.5% likelihood of seeing at least 1 objective tumor response assuming a true ORR of 20%. Patients who do not achieve at least an unconfirmed response within 9 months (must be subsequently confirmed) will be considered non-responders for purposes of this analysis.
Progression-free survival time | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibran Ahmed, Principal Investigator — National Cancer Institute LAO
Locations (3):
- United States (3):
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT05715281/ICF_000.pdf